CLINICAL TRIAL: NCT00685581
Title: Rationale, Study Design and Baseline Data of the TRANSQUAL Clinical Trial: A Study to Evaluate the Impact of Different Milk Fatty Acid Profiles on Cardiovascular Risk Factors in Healthy Volunteers; Focus on Trans Fatty Acids
Brief Title: Impact of Vaccenic Acid Consumption on the Metabolism of Saturated Fatty Acids: Relationship With Cardiovascular Risk Factors
Acronym: TRANSQUAL WPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AU684
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Cardiovascular Disease
Keywords: TFA; SFA; Clinical trial; fat milk
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): Arms A: the lowest R-TFA/SFA ratio obtained from dairy cows in Winter period
  Interventions: Dietary Supplement: Ruminant trans fatty acid enriched diet - lowest ratio
- B (Experimental): Arms B: the medium R-TFA/SFA ratio obtained from dairy cows feeding with Winter diet supplemented with 4.1% flax seed.
  Interventions: Dietary Supplement: Ruminant trans fatty acid enriched diet - medium ratio
- C (Experimental): Arms C: the highest R-TFA/SFA ratio obtained from dairy cows feeding with Winter diet supplemented with 9% flax seed.
  Interventions: Dietary Supplement: Ruminant trans fatty acid enriched diet - highest ratio

INTERVENTIONS:
Dietary Supplement: Ruminant trans fatty acid enriched diet - lowest ratio — the lowest R-TFA/SFA ratio obtained from dairy cows in Winter period
  Arms: A
Dietary Supplement: Ruminant trans fatty acid enriched diet - medium ratio — the medium R-TFA/SFA ratio obtained from dairy cows feeding with Winter diet supplemented with 4.1% flax seed
  Arms: B
Dietary Supplement: Ruminant trans fatty acid enriched diet - highest ratio — the highest R-TFA/SFA ratio obtained from dairy cows feeding with Winter diet supplemented with 9% flax seed
  Arms: C

SUMMARY:
The investigators' project has for principal objective to evaluate the impact of three specific ruminant milk fats with a Trans Fatty Acid content ranging from 2.9% to 12.2% obtained by modification of the cow's diet on cardiovascular risk factors in healthy subjects.

DETAILED DESCRIPTION:
111 healthy, normolipemic men and women (18y to 50y) have been recruited for a monocentric, randomised, double-blind, controlled 4-week study. All the volunteers consumed 3 experimental products (butter, dessert cream and cakes) made with one of the 3 specific milk fats up to 55 g fat/day.

ELIGIBILITY:
Inclusion Criteria:

* HDL cholesterol, g/L > 0.4
* Triacylglycerol g/L <1.50
* LDL Cholesterol g/L <1.60
* Waist size < 94 cm (men) or 80 cm (women)
* Affiliated to National Health Insurance
* Normal blood pressure (diastolic <90 mm Hg, systolic <140 mm Hg)
* For women: effective contraception
* Subject giving his/her written informed consent
* Subject willing to comply with the study procedures

Exclusion Criteria:

* Reported food allergies
* Currently participating or having participated in another clinical trial during the last 4 weeks prior to the beginning of this study
* Hepatic or renal impairments
* Positive serologies to HIV or HCV,
* Blood donation done less than 2 months before the start of the study
* Chronic pathologies
* Refusal to be registered on the National Volunteers Data file
* Being in exclusion on the National Volunteers Data file

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2007-04; Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
HDL-cholesterol

SECONDARY OUTCOMES:
total cholesterol
LDL-cholesterol
triglycerides
apolipoprotein

CONTACTS AND LOCATIONS:
Overall Officials: Yves Boirie, MD, PhD, PU-PH, Principal Investigator — UMR1019 INRA-Université Clermont1; Jean-Michel Chardigny, PhD, Study Director — UMR1019 INRA-Université Clermont1
Locations (1):
- Centre de Recherche en Nutrition Humaine (CRNH), UEN, Laboratoire de Nutrition Humaine, Clermont-Ferrand, France